CLINICAL TRIAL: NCT03773081
Title: SOLVE-ACS: Prospective Multicenter Evaluation of the Performance of the Bioresorbable Magnesium-Stents Magmaris in Patients With Acute Coronary Syndrome (ACS)
Brief Title: SOLVE-ACS: Bioresorbable Magnesium-Stents Magmaris in ACS Lesions
Acronym: SOLVE-ACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, David Manuel Leistner, Coordinating Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4.1
Record Dates: First submitted 2018-12-09; First posted 2018-12-12 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Acute Coronary Syndrome; STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation MI
Keywords: Acute Coronary Syndrome; STE-ACS; NSTE-ACS; Magmaris
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magmaris implantation (Other): Subjects will undergo a PCI for the implantation of the Magmaris scaffold in accordance with the standard of care and standard hospital practice.
  Interventions: Device: Implantation of the Magmaris scaffold

INTERVENTIONS:
Device: Implantation of the Magmaris scaffold — Subjects will undergo a PCI for the implantation of the Magmaris scaffold in accordance with the standard of care and standard hospital practice. Maximum of one single ACS-causing de novo lesions in one separate major epicardial vessels is allowed.

SUMMARY:
The aim of the registry is to investigate the clinical performance of the Magmaris Magnesium Stent in STE-ACS and NSTE-ACS patients.

DETAILED DESCRIPTION:
The Magmaris Magnesium-Stent is indicated for improving luminal diameter and stabilize culprit lesions in patients with coronary artery disease (CAD) including ST-segment elevation (STE-) as well as Non-ST-segment elevation (NSTE-) acute coronary syndrome (ACS). Patients scheduled for this registry, must have one angiographic clear detectable ACS-causing culprit lesion with a reference diameter and a lesion length, which closely match the nominal Magmaris reference diameter and length.

Primary endpoint will be the procedural angiographical success at the end of PCI, defined as successful Magmaris implantation at the "culprit lesion site" with less than 30% final stenosis (by visual estimation) and distal TIMI 3 flow. Secondary endpoints will include clinical and angiographic parameters as well as parameters gained through OCT-imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of 18 - 70 years of age
* STE- or NSTE-ACS with planned invasive therapy strategy
* At least coronary one-vessel disease with one angiographically detectable "culprit lesion"
* Target lesion length ≤ 21 mm and its diameter is ≥ 2.7mm and ≤ 3.7 mm by QCA or by visual estimation.
* Subject is eligible for Dual Anti Platelet Therapy (DAPT) for 12 months after ACS

Additional inclusion criteria MCG-substudy:

* Hospitalization for NSTE- ACS in low- and/or risk-class (GRACE-Score ≤ 170) with planned invasive therapy

Exclusion Criteria:

* Currently participating within a FIM or RCT and primary endpoint is not reached yet.
* Known allergies to: Acetylsalicylic Acid (ASA), clopidogrel, ticlopidine, prasugrel, heparin or any other anticoagulant /antiplatelet required for PCI, contrast medium, sirolimus, or similar drugs or the Magmaris materials including Magnesium, Yttrium, Neodymium, Zirconium, Gadolinium, Dysprosium, Tantalum that cannot be adequately pre-medicated.
* Renal insufficiency with serum-creatinine ≥ 2.5 mg/dl or subjects on dialysis.
* Known systolic heart failure with left-ventricular ejection fraction (LV-EF≤ 30 %).
* Active sepsis.
* Presence of cardiogenic shock or heart failure requiring intubation, inotropes, intravenous diuretics or mechanical circulation support.
* Refractory ventricular arrhythmia requiring pharmacologic or defibrillator therapy.
* Patients under immunosuppressive therapy.
* Unprotected significant left main- stenosis.
* ACS with culprit lesion in a bypass graft or ACS caused by stent/BVS-thrombosis or stent/BVS-restenosis.
* ACS caused by left main coronary artery disease or an ostial target lesion (within 5.0 mm of vessel origin).
* Culprit lesion involves a side branch ≥2.0 mm in diameter (bifurcation lesion).
* Culprit lesion located within a true vessel bifurcation (including side branch > 2mm) which requires bifurcation-treatment according to the investigator's discretion.
* Extent and severity of CAD is such that investigator believes it is likely that bypass surgery will be required within 1 year of enrollment.
* Severe calcification or extreme tortuosity of vessel with "culprit lesion".
* Culprit lesion with very distal location.
* Culprit vessels with "low or no-reflow phenomenon" (TIMI 0,I,II) after mechanical recanalization or pre-dilatation using a non-compliant balloon with 1:1 balloon-to-artery ratio.
* Culprit lesions with a length ≥ 21 mm or within vessels with reference diameter≤ 2.7mm or ≥ 3.7 mm by QCA or by visual estimation.
* Unsuccessful pre-dilatation, defined as minimal lumen diameter smaller than the respective crossing profile of Magmaris and angiographic complications (e.g. distal embolization, side branch closure, extensive dissections), by visual estimation.

Additional exclusion criteria MCG-substudy:

* Non-MCG-safe metal implants
* Inability or unwillingness to lie flat for 5 minutes and follow breathing commands

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Procedural angiographical success | At the end of PCI
  Procedural angiographical success at the end of PCI, defined as successful Magmaris implantation at the "culprit lesion site" with less than 30% final stenosis (by visual estimation) and distal TIMI 3 flow.

SECONDARY OUTCOMES:
ST-segment resolution at the electrocardiogram (ECG) | Within 60 minutes of primary PCI
  ST-segment resolution at ECG.
Procedural clinical success within hospital stay | Until hospital discharge, an expected average of 4 days
  No in-hospital clinically-driven target lesion revascularization.
Target lesion revascularization | 6 months, 12 months and 2 years
  Clinical driven target-lesion revascularization with the use of either PCI or CABG at 6 months, 12 months and at 2 years follow-up respectively.
Device-oriented composite endpoint (DOCE) | 6 months, 12 months and 2 years
  Device-oriented composite (DOCE) endpoint of cardiac death, target vessel-related reinfarction and ischemia-driven target-lesion revascularization at 6 months, 12 months and at 2 years follow-up respectively.
Major adverse cardiovascular events (MACE) | Until hospital discharge, 6 months, 12 months and 2 years
  Cardiac death, any TV-MI, target vessel revascularization (TVR) in-hospital or during follow-up (6 months, 12 months, 2 years).
All-cause death at all time points | Until hospital discharge, 6 months, 12 months and 2 years
  Clinical Endpoint (in-hospital and at follow-up (6 months, 12 months, 2 years).
Cardiac death at all time points | Until hospital discharge, 6 months, 12 months and 2 years
  Clinical Endpoint (in-hospital and at follow-up (6 months, 12 months, 2 years).
Magmaris Thrombosis | Until hospital discharge, 6 months, 12 months and 2 years
  Any definite/probable per ARC defintion Magmaris thrombosis (in-hospital and during follow-up (6 months, 12 months, 2 years).
Any Bleeding | Until hospital discharge, 6 months, 12 months and 2 years
  Bleedings defined according to the Bleeding Academic Research Consortium (BARC) in-hospital and at follow-up (in-hospital and at follow-up (6 months, 12 months, 2 years).
Vascular cerebral events | Until hospital discharge, 6 months, 12 months and 2 years
  Vascular events documented by neurological permanent disabilities or by diagnostic imaging (MRI or CT) in-hospital and during follow-up (6 months, 12 months, 2 years).
Stable angina | 6 months, 12 months and 2 years
  Angina as assessed by Seattle angina score (SAS) at follow-up (6 months, 12 months, 2 years).
Evidence for myocardial ischemia | 12 months
  Clinical or ECG-signs for myocardial ischemia during exercise ECG at 12-month follow-up.
Percent diameter stenosis | 24 months
  Percent diameter stenosis (%DS) at in in-segment (target lesion), in-device, proximal and distal (initial and in case of clinical-indicated re-angiography) (assessed by outcome-blinded Corelab analyses, Charite).
Minimal Lumen Diameter (MLD) | 24 months
  Minimal Lumen Diameter in-segment (target lesion), in-device, proximal and distal (initial and in case of clinical-indicated re-angiography) (assessed by outcome-blinded Corelab analyses, Charite).
TIMI-flow | 24 month
  TIMI-flow before (after mechanical recanalization) and after Magmaris Implantation (assessed by outcome-blinded Corelab analyses, Charite).
ACS-causing "culprit lesion" (OCT) | 24 months
  Mechanism of ACS (Plaque-Rupture vs. Plaque-Erosion vs. other mechanisms) and culprit-plaque-characteristics (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Max/Mean/minimal Mg-Stent diameter/area after implantation and lumen late loss (OCT) | 24 months
  Max/Mean/minimal Mg-Stent diameter/area after implantation and (in case of any clinical indicated re-angiography) lumen late loss as difference Re-OCT to baseline-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Mean/minimal lumen diameter/area/volume | 24 months
  Mean/minimal lumen diameter/area/volume within the target lesion before and after Magmaris-Implantation, as well as (in case of any clinical indicated re-angiography) as difference Re-OCT to baseline-OCT (after Magmaris Implantation) (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Mean/minimal flow-area/volume | 24 months
  Mean/minimal flow-area/volume as difference Re-OCT to baseline-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Intraluminal defect area/volume | 24 months
  Intraluminal defect area/volume at time point re-angiography/Re-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Modified vascular healing score | 24 months
  Modified vascular healing score (%HS; according to Räber EuroIntervention 2016; Sabate + Joner EHJ 2016) as difference Re-OCT to baseline-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Presence of both malapposed and uncovered struts | 24 months
  Presence of both malapposed and uncovered struts (%MN) of the Mg-stent, which is an individual component of the endpoint "Healing Score" as difference Re-OCT to baseline-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Presence of uncovered struts alone | 24 months
  Presence of both uncovered struts of the Mg-stent, which is an individual component of the endpoint "Healing Score" as difference Re-OCT to baseline-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Presence of malapposed struts alone | 24 months
  Presence of both malapposed struts of the Mg-stent which is an individual component of the endpoint "Healing Score" as difference Re-OCT to baseline-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Incomplete strut apposition (ISA) area/volume | 24 months
  Incomplete strut apposition (ISA) area/volume as difference Re-OCT to baseline-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Percentage of covered struts | 24 months
  Percentage of covered struts at Re-OCT follow-up (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Mean/maximal thickness of the struts coverage | 24 months
  Mean/maximal thickness of the struts coverage at Re-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Neointimal hyperplasia area/volume | 24 months
  Neointimal hyperplasia area/volume at Re-OCT (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Thickness of neointimal tissue developed over lipid rich plaque | 24 months
  Thickness of neointimal tissue developed over lipid rich plaque at Re-OCT follow-up (assessed by outcome-blinded OCT Corelab analyses German Heart Center Munich: Prof. Dr. M. Joner).
Diagnostic accuracy values (sensitivity, specificity, PPV, NPV, positive and likelihood ratios) of MCG determination (MCG-substudy) | 24 months
  Diagnostic accuracy values (sensitivity, specificity, PPV, NPV, positive and likelihood ratios) of MCG determination (ST-T Score (Angle dynamic), ST-T-analysis (distance parameter and rato-dynamics), PLP2 Score, VMCG Score (T-begin till Tmax and RP ½ till Tmax), T-dispersion Score) for the vessel with target lesion compared to angiography at ACS. A comparison to exercise-ECG at 12 months will also be performed.
Diagnostic accuracy values (sensitivity, specificity, PPV, NPV, positive and likelihood ratios) of MCG Determination (MCG-substudy) | 24 months
  Diagnostic accuracy values (sensitivity, specificity, PPV, NPV, positive and likelihood ratios)of MCG determination (ST-T Score (Angle dynamic), ST-T-analysis (distance parameter and rato-dynamics) PLP2 Score, VMCG Score (T-begin till Tmax and RP ½ till Tmax), T-dispersion Score) for characteristics of the ACS-causing "culprit lesion" compared to OCT before Magmaris-Implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Landmesser, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (4):
- Germany (4):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Johannes Wesling, Minden